CLINICAL TRIAL: NCT06261866
Title: Multimodality Imaging and Functional Lesion Assessment in Intermediate Grade Coronary Stenosis in Chronic Coronary Syndrome: MultiInter-CCS Study
Brief Title: Multimodality Imaging and Functional Lesion Assessment in Intermediate Coronary Stenosis in Chronic Coronary Syndrome
Acronym: MultiInter-CCS
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, MD, PhD, FESC, Medical University of Warsaw
Other Study IDs: MultiInter-CCS
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Chronic Coronary Syndrome
Keywords: FFR; OCT; IVUS; CCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic coronary syndromes identified with intermediate grade coronary stenosis: Patients chronic coronary syndrome identified with intermediate grade coronary stenosis undergo coronary angiography according to current practice and guidelines recommendations. FFR will be measured, in consistency with the guidelines and recommended clinical practice. In case of FFR > 0.8 optimal pharmacotherapy will be prescribed; on the contrary, in case of FFR ≤ 0.8 PCI will be performed. OCT imaging will be performed with commercially available device (Abbott, C7XR Dragonfly TM LightLab Imaging Inc., MA, USA) using the non-occlusive flushing technique.

SUMMARY:
The aim of this prospective, investigator-initiated study is to evaluate the diagnostic accuracy and correlations between functional indices (fractional flow reserve, FFR) and morphometric indices: luminal and qualitative parameters assessed by optical coherence tomography (OCT) including minimal lumen area, plaque type, presence of thin cap fibroatheroma among patients with chronic coronary syndrome identified with intermediate grade coronary stenosis.

DETAILED DESCRIPTION:
This is a prospective, single center, non-randomized, single-arm, investigator-initiated study evaluating diagnostic accuracy and correlations between functional indices (fractional flow reserve, FFR) and morphometric indices: luminal and qualitative parameters evaluated by OCT including minimal lumen area, plaque stratification into fibrotic, calcific, lipidic plaque, or thin cap fibroatheroma) among patients with chronic coronary syndrome identified with intermediate grade coronary stenosis.

The additional objectives include: evaluation of the impact of age, sex, diabetes mellitus, renal dysfunction on the assocation between functional and morphometric indices of coronary stenosis.

We hypothesized that in patients with intermediate grade coronary stenosis in chronic coronary syndorme there is a positive correlation between the functional parameters and the morphometric parameters of cornary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Chronic coronary syndrome defined as presence of chest pain ranked 2-3 in the Canadian Cardiovascular Society classification or positive ischemia test (exercise test, single photon emission tomography (SPECT)
* Intermediate grade coronary stenosis of 40-80% assessed visually in coronary angiography
* FFR and OCT examination of the same lesion
* The patient is willing to participate in the study and has provided a written informed consent

Exclusion Criteria:

* Acute coronary syndrome
* Proximal left main lesion
* Ostial right coronary artery lesion
* Bypass of the assessed vessel
* Contraindications for adenosine administration
* Hemodynamic instability
* Heart insufficiency in New York Heart Association (NYHA) class IV scale
* Acute renal insufficiency
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing coronary angiogram due to chronic coronary syndrome with intermediate grade coronary stenosis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between fractional flow reserve (FFR) and minimal lumen area within the coronary stenosis | Baseline
Correlation between fractional flow reserve (FFR) and mean lumen area within the coronary stenosis | Baseline

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Tomaniak, MD, PhD, Assoc. Prof., Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No